CLINICAL TRIAL: NCT06732076
Title: The Effect of a Web-Based Breastfeeding Education Program for Adolescent Pregnant Women in the Third Trimester on Breastfeeding Practices: Randomized Controlled Trial
Brief Title: The Effect of a Web-Based Breastfeeding Education Program for Adolescent Pregnant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Veysel Can, Asst. Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: WEB TABAN
Record Dates: First submitted 2024-11-19; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): web based education
  Interventions: Behavioral: web based education
- control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: web based education — web based education
  Arms: experimental

SUMMARY:
It is crucial to prepare adolescent mothers-who represent a vulnerable group where the importance of breastfeeding is increasingly emphasized-for the breastfeeding process. One potential method for promoting breastfeeding is through web-based education interventions. The aim of this study was to evaluate the effect of a web-based breastfeeding education program, developed by the researchers, on breastfeeding outcomes among adolescent pregnant women in the postpartum period. This randomized controlled study involved a sample of 100 pregnant adolescents, aged 15-19 years, who were in their third trimester of pregnancy. The study commenced after obtaining ethical approval and permissions from the hospital where the research was conducted.

A web-based breastfeeding education program was administered to the experimental group. Data were collected using a Socio-Demographic Data Form, the Breastfeeding Self-Efficacy Scale Short Form (Antenatal Version), the Breastfeeding Self-Efficacy Scale Short Form (Postnatal Version), and the LATCH Breastfeeding Diagnosis and Assessment Scale. Data collection occurred during the third trimester (pretest) and the 1st and 8th postnatal weeks (posttest).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 15 and 19 years
* Had not previously received planned breastfeeding education
* Were between 28 and 37 weeks gestation (third trimester)
* Gave birth at term
* Had no health issues preventing breastfeeding
* Could read, write, and respond to questions
* Had access to a computer, tablet, or smartphone, and had regular internet access.

Exclusion Criteria:

* Participants were excluded if they had multiple pregnancies
* Physical or mental health problems, communication disabilities
* A history of breast surgery
* İf their newborns were considered high-risk.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — adolescent mother
Enrollment: 90 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Breastfeeding self-efficacy scale | pre-test post-test (approximately six month)
  Breastfeeding self-efficacy scale

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Van Yüzüncü Yıl University, Van, Tuşba
  - Van Yüzüncü Yıl University, Van

IPD SHARING:
Plan to Share IPD: No